CLINICAL TRIAL: NCT01321788
Title: Venous Thromboembolism Prophylaxis Post Cesarean Section(PRO-CS-Trial)
Brief Title: Venous Thromboembolism Prophylaxis Post Cesarean Section
Acronym: PROCS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Saud University (Other)
Collaborators: King AbdulAziz City for Science and Technology (Other)
Responsible Party: Principal Investigator, Farjah Hassan AlGahtani, Dr., King Saud University
Other Study IDs: PRO-CS TRIAL
Record Dates: First submitted 2011-03-22; First posted 2011-03-24 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Bleeding; Venous Thromboembolism
Keywords: thromboprophylaxis; pregnancy; post-cesarian section
MeSH Terms: conditions — Hemorrhage; Venous Thromboembolism | interventions — Tinzaparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- STUDY GROUP: will receive the study drug Innohep ® for 14 days
  Interventions: Drug: TINZAPARIN
- CONTROL: The group that will receive placebo for 14 days
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: TINZAPARIN — Eligible women following cesarean section will randomly receive once-daily injections of study drug (4,500 IU tinzaparin sodium within 12 to 24 hours postpartum and continued for two (2) weeks postpartum.
  Other Names: Innohep
  Groups: STUDY GROUP
Drug: PLACEBO — Eligible women following cesarean section will receive a once-daily injections of placebo within 12 to 24 hours postpartum and continued for two (2) weeks postpartum.
  Groups: CONTROL

SUMMARY:
Pregnancy is associated with an overall 5-10 fold increased risk of venous thromboembolism (VTE). VTE remains the most common cause of maternal death in the developed world. It is up to 10 times more common in pregnant women than non-pregnant women of comparable age. More than a third of pregnancy-related VTE occurs during the six weeks after delivery. When compared with vaginal delivery, cesarean delivery further increases the risk of pregnancy associated VTE by three-fold.

DETAILED DESCRIPTION:
This is a double blind- a randomized controlled study of prophylactic LMWH in women at low risk for VTE following a cesarean section procedure. The sample size is 300 patients, Eligible, consenting, and randomized participants will receive once-daily injections of study drug (4,500 IU Tinzaparin Sodium [Innohep®] within 12- to 24-hours postpartum and continue for two weeks versus Placebo in the other arm and follow for six (6) weeks postpartum.

On the day of hospital discharge, bilateral leg imaging with compression, leg ultrasounds, and pelvic vein imaging with MRV will be completed. The primary outcome will be adjudicated, while DVT will be documented on ultrasounds or MRV on the day of hospital discharge. Secondary outcomes will include symptomatic DVT and PE, death from PE, major and minor bleeding, and HIT during the six-week postpartum period. All outcomes will be adjudicated by an independent committee of experts blinded to study drug allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old.
2. Delivered by cesarean section (emergency or planned).
3. Signed, informed consent.
4. Ready access to a local health service.
5. Capable of using Tinzaparin.

Exclusion Criteria:

1. at high risk for thromboembolism (any one of the following):

   * age more than 35 years old
   * obesity (more than 80 kg)
   * parity more than 4
   * gross varicose veins
   * current infection
   * pre-eclampsia
   * immobility prior to surgery (more than 4 days)
   * Major current disease: including heart or lung disease, cancer,inflammatory bowel disease and nephrotic syndrome.
   * Extended major pelvic or abdominal surgery (e.g. cesarean hysterectomy)
   * Patients with a family history of VTE
   * History of superficial phlebitis
2. More than 36 hours since delivery
3. Need for anticoagulation, including:

   * women with a confirmed thrombophilia
   * women with paralysis of lower limbs
   * women with personal history of VTE
   * women with antiphospholipid antibody syndrome (APLA)
   * women with mechanical heart valves
4. Contraindication to heparin therapy, including history of heparin induced thrombocytopenia.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Consecutive adult patients (aged over 18 years) that had been delivered by emergency or elective cesarean section with no previous history of VTE are eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Deep Vein Thrombosis | 24 months
  The primary outcome will be adjudicated, while DVT will be documented on ultrasounds or MRV on the day of hospital discharge.

SECONDARY OUTCOMES:
symptomatic DVT and bleeding | Symptomatic DVT
  . Secondary outcomes will include symptomatic DVT and PE, death from PE, major and minor bleeding, and HIT during the six-week postpartum period.

CONTACTS AND LOCATIONS:
Overall Officials: FARJAH H ALGAHTANI, MD, Principal Investigator — King Saud University
Locations (1):
- Security Forces Hospital, Riyadh, Riyadh Region, Saudi Arabia

REFERENCES:
- [Background] Kujovich JL. Hormones and pregnancy: thromboembolic risks for women. Br J Haematol. 2004 Aug;126(4):443-54. doi: 10.1111/j.1365-2141.2004.05041.x. PMID 15287937
- [Background] Samuelsson E, Hellgren M, Hogberg U. Pregnancy-related deaths due to pulmonary embolism in Sweden. Acta Obstet Gynecol Scand. 2007;86(4):435-43. doi: 10.1080/00016340701207500. PMID 17486465
- [Background] Morris JM, Algert CS, Roberts CL. Incidence and risk factors for pulmonary embolism in the postpartum period. J Thromb Haemost. 2010 May;8(5):998-1003. doi: 10.1111/j.1538-7836.2010.03794.x. Epub 2010 Feb 1. PMID 20128859
- [Background] Chan WS. Venous thromboembolism in pregnancy. Expert Rev Cardiovasc Ther. 2010 Dec;8(12):1731-40. doi: 10.1586/erc.10.169. PMID 21108555
- [Derived] Middleton P, Shepherd E, Gomersall JC. Venous thromboembolism prophylaxis for women at risk during pregnancy and the early postnatal period. Cochrane Database Syst Rev. 2021 Mar 29;3(3):CD001689. doi: 10.1002/14651858.CD001689.pub4. PMID 33779986
- See also: Venous Thromboembolism During Pregnancy — http://www.aafp.org
- See also: Venous Thromboembolism in Pregnancy Study — http://clinicaltrials.gov/ct2/show/NCT00856076
- See also: National Guideline Clearinghouse | Venous thromboembolism — http://www.guideline.gov/content.aspx?id=12966
- See also: Venous thromboembolism in pregnancy — http://www.ncbi.nlm.nih.gov/pubmed/19228606